CLINICAL TRIAL: NCT05861375
Title: Assessment of Liver Damage Using the Fibroscan in Patients With Anorexia Nervosa
Brief Title: Liver Biomarkers in Anorexia Nervosa
Acronym: LIBAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0049
Record Dates: First submitted 2023-02-07; First posted 2023-05-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Anorexia Nervosa
Keywords: Liver Fibrosis; Liver Steatosis; Enteral Refeeding; Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — These are blood samples that may be used for further research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non applicable (NA): Patients with Anorexia Nervosa hospitalized for malnutrition
  Interventions: Diagnostic Test: Fibroscan

INTERVENTIONS:
Diagnostic Test: Fibroscan — Fibroscan is a non-invasive device that allows liver exploration painlessly, quickly (a few minutes) and with immediate results. A probe placed on the skin generates an elastic wave completely painlessly and the device measures its speed of propagation in the liver. Liver stiffness is calculated from this speed.

SUMMARY:
The main goal of the Liver Biomarkers in Anorexia Nervosa (LIBAN) study is to determine the prevalence of liver fibrosis in patient with Anorexia Nervosa.

DETAILED DESCRIPTION:
Prevalence of hepatic fibrosis will be non-invasively investigated, in the Anorexia Nervosa inpatient population, using the Fibroscan ®. Furthermore, liver blood markers will be assessed.

ELIGIBILITY:
Inclusion Criteria :

* Patient over 15 years old
* Diagnosis of Restricted Eating Disorders including Anorexia Nervosa according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Admission to the endocrinology, diabetology and nutrition department of the Nantes University Hospital.

Exclusion Criteria :

* Chronic active viral hepatitis
* Hemochromatosis
* Other genetic, autoimmune, toxic or drug-induced hepatitis
* Treatment with a drug known to induce fatty liver disease (amiodarone, carbamazepine, tamoxifen, valproate, clozapine, anti-retrovirals) unless the dose has been stable for ≥ 3 months
* Excessive alcohol consumption (≥ 30 grams per day in men, ≥ 20 grams per day in women)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive inclusion of patients hospitalized in the endocrinology department for anorexia nervosa with malnutrition criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Liver fibrosis prevalence in patients with Anorexia nervosa | Day one
  Liver stiffness will be assessed using Fibroscan (kPA) within the 24 hours following admission to the endocrinology, diabetology and nutrition department.

CONTACTS AND LOCATIONS:
Overall Officials: Sarra SMATI-GRANGEON, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided